CLINICAL TRIAL: NCT00254956
Title: A Multi-Center, Multinational, Randomized, Double-Blind, Parallel Group Study of the Effects of Ciclesonide Hfa-Mdi 640 μg/Day and Beclomethasone Hfa-Mdi 640 μg/Day on Lens Opacification in Adult Subjects With Moderate to Severe Persistent Asthma
Brief Title: Effects Of Ciclesonide And Beclomethasone On Lens Opacification In Adult Subjects With Moderate To Severe Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Takeda (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SFY6160
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Respiratory Tract Diseases; Respiratory Hypersensitivity; Asthma
Keywords: Diseases; respiratory tract diseases; respiratory hypersensitivity; asthma
MeSH Terms: conditions — Respiratory Tract Diseases; Respiratory Hypersensitivity; Asthma; Disease | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: ciclesonide (XRP1526)

SUMMARY:
The primary objective is to demonstrate the non-inferiority of ciclesonide compared to beclomethasone-HFA in the occurrence of Class 1 lens event for nuclear (NO), cortical (C), or posterior subcapsular (P) lens opacification within 12 months. Secondary objectives are to compare ciclesonide and beclomethasone with respect to class II and class III best corrected visual acuity and intraocular pressure from baseline to 12 months.

DETAILED DESCRIPTION:
This is a multi-center, multinational, active-controlled, double-blind, randomized (1:1) parallel group study of the effects of inhaled ciclesonide HFA-MDI 640 mcg/day and beclomethasone HFA-MDI 640 mcg/day on lens opacification in adult subjects with moderate to severe persistent asthma. The study consists of a 1-14 day screening phase during which subject eligibility will be determined, followed by a 12-month double-blind treatment phase. Lens opacification will be evaluated by slit lamp examination performed after pupillary dilation to at least 6.0 mm before randomization and after 4 months, 8 months, and 12 months of treatment using the LOCS III system for grading lens opacities. Best-corrected visual acuity and intraocular pressure will be measured at each eye examination visit. An Independent Data Monitoring Committee (IDMC) will be constituted to monitor safety throughout the double-blind treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-lactating females 18 years of age and older with a history of moderate to severe persistent asthma for a duration of at least 2 months prior to screening.
* At screening, FEV1 must be ≥ 40% and ≤ 85% of predicted.
* Documented use of inhaled corticosteroid therapy at any dose for at least 1 month prior to screening.
* Able to demonstrate acceptable oral inhaler technique.
* Non-smoker for at least the past year and less than a 10 pack-year smoking history if previous smoker.
* Written informed consent agreement.

Exclusion Criteria:

* History of prior cataract surgery in either eye.
* Evidence of congenital cortical cataract.
* Inability to grade nuclear, cortical, or posterior subcapsular opacities in either eye with LOCS III at the baseline slit lamp examination.
* Inability to dilate pupils to at least 6.0 mm.
* Nuclear opalescence with a LOCS III grade ≥ 4 in either eye at the baseline slit lamp examination.
* Cortical lens opacities with a LOCS III grade ≥ 3 in either eye at the baseline slit lamp examination.
* Posterior subcapsular lens opacities with a LOCS III grade ≥ 2 in either eye at the baseline slit lamp examination.
* Elevated intraocular pressure requiring treatment
* Best corrected visual acuity less than 74 letters (equivalent to vision worse than 20/30) in either eye at baseline.
* Females who are pregnant or lactating or have a positive pregnancy test at Visit 1 (Screening).
* Have had more than 1 in-patient hospitalization in the past year for asthma exacerbations.
* Have had more than 2 bursts of oral steroids per year for each of the past 2 years prior to screening.
* Chronic use of oral, injectable, or topical steroids except for inhaled corticosteroids for any condition. Topical corticosteroids designated as having a mild potency by the Stoughton-Cornell Scale or the European Guideline for levels of corticosteroid activity are allowed (see AppendixG).
* Any chronic condition that is likely to require treatment with oral or systemic corticosteroids other than asthma (e.g. systemic lupus, inflammatory bowel disease, rheumatoid arthritis).
* Topical ocular steroid treatment within 3 months prior to screening.
* Chronic or recurrent inflammatory disease in either eye likely to result in visual abnormalities or require treatment with ocular steroids.
* History of drug or alcohol abuse.
* Any clinically significant medical condition that would interfere with the subject's ability to participate in and comply with study protocol.
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Hypersensitivity to the investigational products or to drugs with similar chemical structures.
* Have been treated with any investigational drug/product within 30 days prior to Visit 1 (Screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1568 (Actual)
Dates: Start 2004-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the occurrence of a Class I lens event for nuclear (NO), cortical (C), or posterior subcapsular (P) lens opacification within 12 months.
A Class I lens event is defined as any of the following events in either eye:
- 1.Increase from baseline in LOCS III grade of ≥ 0.5 (NO), ≥ 0.8 (C), or ≥ 0.5 (P)
- 2.Cataract surgery

SECONDARY OUTCOMES:
- 1.Change from baseline to Month 12 in LOCS III grade for (a) nuclear opalescence, (b) cortical opacity, and (c) posterior subcapsular opacity.
- 2.Occurrence within 12 months in either eye of a Class II lens event: Increase from baseline in LOCS III grade of ≥ 0.9 (NO), ≥ 1.5 (C), or ≥ 0.9 (P), or cataract surgery.
- 3.Occurrence within 12 months in either eye of a Class III lens event: LOCS III grade ≥ 2.0 for any type of opacity (NO, C, or P) and a change in LOCS III grade of ≥ 0.9 for NO, ≥ 1.5 for C, and ≥ 0.9 for P, or cataract surgery.
- 4.Change from baseline to Month 12 in best-corrected visual acuity.
- 5.Change from baseline to Month 12 in intraocular pressure (mm Hg).
Tertiary endpoint:
- Change in post-bronchodilator FEV1 from baseline to Month 12.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Chilly-Mazarin, France

REFERENCES:
- [Derived] Chylack LT Jr, Gross GN, Pedinoff A; Ciclesonide Lenticular Safety Study Group. A randomized, controlled trial to investigate the effect of ciclesonide and beclomethasone dipropionate on eye lens opacity. J Asthma. 2008 Dec;45(10):893-902. doi: 10.1080/02770900802353636. PMID 19085579